CLINICAL TRIAL: NCT04462146
Title: Internet-based Self Applied Treatment Program for Prolonged Grief Disorder (PGD): An Open Clinical Trial
Brief Title: An Internet-based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
Acronym: GROw
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: z7dqxrg8
Record Dates: First submitted 2020-06-17; First posted 2020-07-08 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Prolonged Grief Disorder
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based intervention (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention.
  Interventions: Behavioral: Internet-based Self Applied Treatment Program
- Face-to-face treatment by videoconference (Active Comparator): Face-to-face Intervention by videoconference applied by a therapist: Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention.
  Interventions: Behavioral: Videoconference treatment with a therapist

INTERVENTIONS:
Behavioral: Internet-based Self Applied Treatment Program — It is a self-applied treatment for PGD through the web "psicologíaytecnología.labpsitec.es". There are 8 treatment modules. Each module lasts approximately 60 minutes. It contains written information, videos, audios, photos and interactive questionnaires. The total duration of treatment is up to 8-10 weeks. A weekly support call will be made (maximum 10 minutes) to answer questions and reinforce and motivate the patient. No additional clinical content or counselling will be provided. Main components of the treatment: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Other Names: GROw
  Arms: Internet-based intervention
Behavioral: Videoconference treatment with a therapist — It is a treatment for PGD applied by a therapist composed of 8-10 treatment sessions. Each session lasts approximately 60 minutes. No weekly support call will be provided.
  The sessions will take place by videoconference. Main components of the treatment: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention.
  Arms: Face-to-face treatment by videoconference

SUMMARY:
The purpose of this study is to investigate the feasibility, acceptability and preliminary efficacy of an internet delivered cognitive behavior treatment (ICBT) for people with prolonged grief disorder (PGD) compared to a face-to-face intervention for PGD.

DETAILED DESCRIPTION:
Grief is an intense emotional reaction to the loss of a loved one. It produces feelings of regret and longing that usually decrease over time. However, some people have difficulty adapting to the loss and develop Prolonged Grief Disorder (PGD). An open clinical trial will be conducted to investigate the feasibility [initial efficacy and acceptability] of an Internet delivered cognitive behavior treatment (ICBT) for adult people diagnosed with prolonged grief disorder (PGD). There will be at least 24 participants that will be randomly assigned to experimental group (internet-based treatment for PGD) or active control group (traditional face- to-face intervention for PGD). Four assessment moments will be included (pre-treatment, post-treatment, 3 months follow-up and 12 months follow-up). The present study aims to improve knowledge about the feasibility, acceptability and preliminary efficacy of an ICBT for PGD and conduct a preliminary comparison between two intervention conditions (internet-based intervention vs. traditional face-to-face intervention). Also, the investigators aim to collect information that can help to improve the efficacy and acceptability of Internet-based interventions in general.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Meeting diagnostic criteria for PGD
* Sign an informed consent
* Ability to understand and read Spanish
* Ability to use a computer and having access to the Internet
* Having an e-mail address

Exclusion Criteria:

* Presence of risk of suicide or self-destructive behaviors
* Presence of another severe mental disorder (substance abuse or dependence, psychotic disorder, dementia o bipolar disorder)
* Presence of severe personality disorder
* Presence of a medical condition whose severity or characteristics prevent the performance of treatment
* Receiving other psychological treatment during the study for PGD
* An increase and/or change in the medication during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Inventory of Complicated Grief (ICG) validated in the Spanish population | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument that assesses grief symptoms in adults. Good psychometric properties; cronbach's alpha of0.94 in the original version and 0.88 in the Spanish adaptation.
  It consists of 19 items with five response categories (Likert): 0; never 1; rarely 2; sometimes 3; often and 4; forever. The items value the frequency of the symptom explored (emotional, cognitive or behavioral). It is completed in approximately 10 minutes.
  The total score is calculated by adding the score of the 19 items. The total score ranges from 0 to 76, with highest scores corresponding to a greater probability of suffering complicated grief.
Change in the Beck Depression Inventory - Second Edition validated in the Spanish population | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument that assesses characteristic attitudes and symptoms of depression. Psychometric properties; Cronbach's alpha of 0.76 to 0.95 and test-retest reliability of around 0.8. It consists of 21 items that are scored on a scale from 0 to 3. It is calculated by adding the score of the 21 items and the maximum total score is 63.

SECONDARY OUTCOMES:
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) validated in the Spanish population | immediately pre-treatment, weekly during treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess the frequency and severity of anxiety. It also measures the level of avoidance, work, academic, and home interference, and social interference associated with anxiety. Psychometric properties; Cronbach's alpha of 0.80 in the original version and 0.86 in the Spanish adaptation. It consists of 5 items that are scored on a scale of 0 to 4. It is calculated by adding the score of the 5 items and the maximum score is 20.
Change in the Overall Depression Severity and Impairment Scale (ODSIS) validated in the Spanish population | immediately pre-treatment, weekly during treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess the frequency and severity of depression. It also measures the level of avoidance, work, academic, and home interference, and social interference associated with depression. Psychometric properties; Cronbach's alpha of 0.91 to 0.94 in the original version and good convergent and discriminant validity.
  Cronbach's alpha of 0.93 in the Spanish adaptation and excellent convergent and discriminant validity. It consists of 5 items that are scored on a scale of 0 to 4. It is calculated by adding the score of the 5 items and the maximum score is 20.
Change in the Positive and Negative Affect Schedule (PANAS) validated in the Spanish population | immediately pre-treatment, weekly during treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess two independent dimensions of affectivity: Positive Affect (PA) and Negative Affect (NA). Psychometric properties; excellent internal consistency in the original version (α = 0.84 to 0.90) and convergent and discriminant validity. Excellent internal consistency in the Spanish adaptation (α =0.87 to 0.91). It consists of 20 items that are scored on a 1-5 scale. It has two subscales: positive affect (10 items) and negative affect (10 items). It is calculated by adding each of the items on the two scales separately. The maximum score is 50 for each of the subscales.
Change in the Quality of Life Index (QLI) validated in Spanish language | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess health-rated quality of life. Psychometric properties; high test-retest reliability (r = .87) and internal consistency (α = .92) in the original version and good test-retest reliability and internal consistency (α = 0.87) in the Spanish language adaptation. It consists of 10 items that assess a global perception of quality of life and aspects ranging from physical well-being to spiritual fulfillment. A 10-point Likert scale is used to measure satisfaction in each area.
Change in the Work and Social Adjustment Scale (WSAS) validated in Spanish language | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess psychosocial functional impairment. Psychometric properties; good to excellent test-retest reliability, sensitivity to change and internal consistency (α = 0.70 to 0.94) in the original version. Good concurrent validity and excellent internal consistency in the Spanish version. It consists of 5 items that are scored on a scale of 0 (not at all) to 8 (very severely). It is calculated adding the score of all the items and the maximum total score is 40. Higher scores indicate greater interference in different areas.
Change in the Posttraumatic Growth Inventory (PTGI) validated in Spanish language | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess post-trauma growth and self-improvement. Psychometric properties; excellent internal consistency (α = 0.90) and acceptable test-retest reliability (around 0.71) in the original version and excellent internal consistency (α = 0.92) in the Spanish version. Is a 21-item scale built on the five-factor model (Factors: Relating to Others, New Possibilities, Personal Strength, Spiritual Enhancement, Appreciation). A 6-point likert scale is used for each item. A summation of the scores indicates the level of post-traumatic growth. Higher score indicates greater positive transformation.
Change in Five-Facet Mindfulness Questionnaire (FFMQ-15) validated in Spanish population | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a short form of the 39-item FFMQ (Baer et al., 2006), self-applied instrument to assess the ability to be aware in the experience of the moment.
  It is a 15-item scale with a Likert response format ranging from 1 (never or very rarely true) to 5 (very often or always true). It evaluates five facets of mindfulness (Observing, Describing, Acting with awareness, Non judging internal experience, Non reactivity to internal experience). Higher scores represent higher dispositional mindfulness.
  Psychometric properties; Good internal consistency is shown on all 5 scales.
Change in Self-Compassion Scale Short Form (SCS-SF) validated in Spanish population | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess the capacity for self-compassion. Psychometric properties; good internal consistency (α = 0.86) and high correlation with the long version of the SCS (r = 0.97) in the original validation and good internal consistency (α = 0.85) and high test-retest reliability in the Spanish version.
  To calculate the total self-compassion score, a total mean is calculated considering the inverse items. Subscale scores are computed by calculating the mean of subscale item responses.
Change in Typical Beliefs Questionnaire (TBQ) | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess maladaptive thinking common in people with complicated grief. Psychometric properties; good internal consistency for the general scale (α = 0.83) and good test-retest reliability.
  Ii is a 25-item scale which measures the degree of agreement regarding different statements with a Likert response format ranging from 0 (not at all) to 4 (very strongly). Five-factor structure (protesting the death, negative thoughts about the world, needing the person, less grief is wrong and grieving too much). The maximum score is 100. The scores of the subscale are obtained from the sum of the elements of each factor.
Change in Purpose-In-Life Test (PIL- 10) | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a short form of the 20-items Purpose-In-Life Test (Crumbaugh, 1968). Is a self-applied instrument to assess the personal experience of meaning of life (satisfaction and meaning of life and vital goals and purposes).
  Psychometric properties; good internal consistency (α = 0.86). The total score is obtained by adding the values of the selected answer options and the maximum score is 70. Two- factor structure (satisfaction and meaning of life; vital goals and purposes).

OTHER OUTCOMES:
Change in Prolonged Grief Disorder-13 (PG-13) validated in Spanish population | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is a self-applied instrument to assess prolonged grief in people who have lost a loved one six or more months ago.
  Psychometric properties; reliability test-retest Kappa coefficient = 1 and Cronbach's alpha = 0.92 in the Spanish adaptation.
  13-item scale grouped into 5 criteria (loss of a loved one, symptoms of intense separation anxiety, duration, cognitive, emotional or behavioral symptoms and functional impairment). Items valued differently according to criteria; Likert-type scale of five responses from 1 (absence of that symptom) to 5 (highest intensity) and dichotomous answer (yes / no). Needed to meet the five criteria to consider prolonged grief.
Change in ADIS Clinician's severity rating scale | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  Indicate the level of distress-interference in functioning. 1 item (from 0/"Absent" to 8/"Very severely disturbing/ disabling") assessed by the therapist.
Change in The Structured Clinical Interview for Complicated Grief (SCI-CG) | immediately pre-treatment, immediately post-treatment, 3-month post-treatment, 12-month post-treatment
  It is an interview with 31 items that evaluates symptoms of prolonged grief in people who have lost a loved one six or more months ago the interview.
  Psychometric properties; acceptable internal consistency (α = 0.86) excellent inter-rater reliability and good test-retest reliability.
  Each item is answered on a 3-point likert scale (Not present, insecure or misleading and present). It is calculated by adding the scores of each item and the highest score is 93.
Change in Expectations and satisfaction Questionnaire | immediately pre-treatment, immediately post-treatment
  It is a self-applied instrument Adapted from Borkovec & Nau (1972) to assess participants' expectations (before the intervention) and satisfaction with the treatment (after the intervention).
  Evaluates the logic of the intervention, satisfaction with the intervention, recommendation of the intervention to others, utility of the intervention for other psychological problems, utility of the intervention for that condition and aversion generated by the intervention. Items are scored on 0-10 scales (0 ="not at all"; 10 = "a lot"). Higher score indicates greater expectation towards treatment and satisfaction with the intervention.
Qualitative opinion interview | immediately post-treatment
  * Perceived clinical utility of each part of the treatment (0 = no useful at all; 10 = maximum utility)
  * Utility images, video, audio and written content (0 = no useful at all; 10 = maximum utility)
  * Utility, satisfaction and help in the adherence of the weekly call (only in internet-based condition group)
Preference scale | immediately pre-treatment, immediately post-treatment
  It is a 7-item scale developed specifically for this study, which evaluates the preferences of the participants on the two treatment conditions (face-to-face and internet-based intervention).
  The 7 items measure general preference, utility, logic and aversiveness of the treatment and recommendation of the intervention to others. The answer to each item is dichotomous: A) self-applied via the Internet (with a short weekly phone call from a therapist); B) Applied weekly face-to-face sessions of approximately 60 minutes, and carried out by a therapist.
Usability and Acceptance Questionnaire | immediately post-treatment
  It is a 11-item questionnaire to assess the usability and acceptance of the technology by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, psychology, Study Director — Universitat Jaume I; Daniel Campos, psychology, Study Director — Universitat Jaume I; Cintia Tur, psychology, Study Chair — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauro C, Reynolds CF, Maercker A, Skritskaya N, Simon N, Zisook S, Lebowitz B, Cozza SJ, Shear MK. Prolonged grief disorder: clinical utility of ICD-11 diagnostic guidelines. Psychol Med. 2019 Apr;49(5):861-867. doi: 10.1017/S0033291718001563. Epub 2018 Jun 18. PMID 29909789
- [Background] Prigerson HG, Horowitz MJ, Jacobs SC, Parkes CM, Aslan M, Goodkin K, Raphael B, Marwit SJ, Wortman C, Neimeyer RA, Bonanno GA, Block SD, Kissane D, Boelen P, Maercker A, Litz BT, Johnson JG, First MB, Maciejewski PK. Prolonged grief disorder: Psychometric validation of criteria proposed for DSM-V and ICD-11. PLoS Med. 2009 Aug;6(8):e1000121. doi: 10.1371/journal.pmed.1000121. Epub 2009 Aug 4. PMID 19652695
- [Background] Estevan, P., del Miguel, C., Prigerson, H., García-García, JA., del Cura, & GEDUPROL. (2019). Adaptación trascultural y validación del cuestionario PG-13 para la detección precoz de duelo prolongado. Psicooncología, 14(1), 163-164. https://doi.org/10.5209/PSIC.55820
- [Background] Bui E, Mauro C, Robinaugh DJ, Skritskaya NA, Wang Y, Gribbin C, Ghesquiere A, Horenstein A, Duan N, Reynolds C, Zisook S, Simon NM, Shear MK. THE STRUCTURED CLINICAL INTERVIEW FOR COMPLICATED GRIEF: RELIABILITY, VALIDITY, AND EXPLORATORY FACTOR ANALYSIS. Depress Anxiety. 2015 Jul;32(7):485-92. doi: 10.1002/da.22385. Epub 2015 Jun 9. PMID 26061724
- [Background] Prigerson HG, Maciejewski PK, Reynolds CF 3rd, Bierhals AJ, Newsom JT, Fasiczka A, Frank E, Doman J, Miller M. Inventory of Complicated Grief: a scale to measure maladaptive symptoms of loss. Psychiatry Res. 1995 Nov 29;59(1-2):65-79. doi: 10.1016/0165-1781(95)02757-2. PMID 8771222
- [Background] Limonero Garcia, J., Lacasta Reverte, M., Garcia Garcia, J., Mate Mendez, J., & Prigerson, H. (2009). Adaptación al castellano del inventario de duelo complicado. Medicina Paliativa, 16(5), 291-297.
- [Background] Beck, A.T., Steer, R.A., y Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] Sanz, J., Navarro, M. E., y Vázquez, C. (2003). Adaptación española del Inventario para la Depresión de Beck-II (BDI-II): 1. Propiedades psicométricas en estudiantes universitarios. Análisis y Modificación de Conducta, 29, 239-288.
- [Background] Campbell-Sills L, Norman SB, Craske MG, Sullivan G, Lang AJ, Chavira DA, Bystritsky A, Sherbourne C, Roy-Byrne P, Stein MB. Validation of a brief measure of anxiety-related severity and impairment: the Overall Anxiety Severity and Impairment Scale (OASIS). J Affect Disord. 2009 Jan;112(1-3):92-101. doi: 10.1016/j.jad.2008.03.014. Epub 2008 May 16. PMID 18486238
- [Background] Gonzalez-Robles A, Mira A, Miguel C, Molinari G, Diaz-Garcia A, Garcia-Palacios A, Breton-Lopez JM, Quero S, Banos RM, Botella C. A brief online transdiagnostic measure: Psychometric properties of the Overall Anxiety Severity and Impairment Scale (OASIS) among Spanish patients with emotional disorders. PLoS One. 2018 Nov 1;13(11):e0206516. doi: 10.1371/journal.pone.0206516. eCollection 2018. PMID 30383797
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Mira A, Gonzalez-Robles A, Molinari G, Miguel C, Diaz-Garcia A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos R, Botella C. Capturing the Severity and Impairment Associated With Depression: The Overall Depression Severity and Impairment Scale (ODSIS) Validation in a Spanish Clinical Sample. Front Psychiatry. 2019 Apr 9;10:180. doi: 10.3389/fpsyt.2019.00180. eCollection 2019. PMID 31024352
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Diaz-Garcia A, Gonzalez-Robles A, Mor S, Mira A, Quero S, Garcia-Palacios A, Banos RM, Botella C. Positive and Negative Affect Schedule (PANAS): psychometric properties of the online Spanish version in a clinical sample with emotional disorders. BMC Psychiatry. 2020 Feb 10;20(1):56. doi: 10.1186/s12888-020-2472-1. PMID 32039720
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Weiss, T., & Berger, R. (2006). Reliability and validity of a Spanish version of the posttraumatic growth inventory. Research on Social Work Practice, 16(2), 191-199. https://doi.org/10.1177/1049731505281374
- [Background] Mezzich, J. E., Cohen, N. L., & Ruiperez, M. A. (1996). A Quality of Life Index: Brief description and validation. Paper presented at the International Congress of the International Federation for Psychiatric Epidemiology. Santiago de Compostela, Spain.
- [Background] Mezzich JE, Ruiperez MA, Perez C, Yoon G, Liu J, Mahmud S. The Spanish version of the quality of life index: presentation and validation. J Nerv Ment Dis. 2000 May;188(5):301-5. doi: 10.1097/00005053-200005000-00008. PMID 10830568
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Echezarraga A, Calvete E, Las Hayas C. Validation of the Spanish Version of the Work and Social Adjustment Scale in a Sample of Individuals With Bipolar Disorder. J Psychosoc Nurs Ment Health Serv. 2019 May 1;57(5):44-51. doi: 10.3928/02793695-20181128-02. Epub 2018 Dec 4. PMID 30508459
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Asensio-Martinez A, Masluk B, Montero-Marin J, Olivan-Blazquez B, Navarro-Gil MT, Garcia-Campayo J, Magallon-Botaya R. Validation of Five Facets Mindfulness Questionnaire - Short form, in Spanish, general health care services patients sample: Prediction of depression through mindfulness scale. PLoS One. 2019 Apr 2;14(4):e0214503. doi: 10.1371/journal.pone.0214503. eCollection 2019. PMID 30939151
- [Background] Garcia-Campayo J, Navarro-Gil M, Andres E, Montero-Marin J, Lopez-Artal L, Demarzo MM. Validation of the Spanish versions of the long (26 items) and short (12 items) forms of the Self-Compassion Scale (SCS). Health Qual Life Outcomes. 2014 Jan 10;12:4. doi: 10.1186/1477-7525-12-4. PMID 24410742
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Skritskaya NA, Mauro C, Olonoff M, Qiu X, Duncan S, Wang Y, Duan N, Lebowitz B, Reynolds CF 3rd, Simon NM, Zisook S, Shear MK. Measuring Maladaptive Cognitions in Complicated Grief: Introducing the Typical Beliefs Questionnaire. Am J Geriatr Psychiatry. 2017 May;25(5):541-550. doi: 10.1016/j.jagp.2016.09.003. Epub 2016 Sep 19. PMID 27793576
- [Background] García-Alandete, J., Martínez, E. R., & Nohales, P. S. (2013). Estructura factorial y consistencia interna de una versión española del Purpose-In-Life Test. Universitas Psychologica, 12(2), 517-530. https://doi.org/10.11144/Javeriana.UPSY12-2.efci
- [Background] Crumbaugh JC. Cross-validation of Purpose-in-Life test based on Frankl's concepts. J Individ Psychol. 1968 May;24(1):74-81. No abstract available. PMID 4385494
- [Derived] Tur C, Campos D, Herrero R, Mor S, Lopez-Montoyo A, Castilla D, Quero S. Internet-delivered Cognitive-Behavioral Therapy (iCBT) for Adults with Prolonged Grief Disorder (PGD): A Study Protocol for a Randomized Feasibility Trial. BMJ Open. 2021 Jul 6;11(7):e046477. doi: 10.1136/bmjopen-2020-046477. PMID 34230018
- See also: International Classification of Diseases 11th Revision — https://icd.who.int/browse11/l-m/en